CLINICAL TRIAL: NCT03580343
Title: Tofacitinib for the Treatment of Inflammatory Eye Disease
Brief Title: Tofacitinib for Inflammatory Eye Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tofacitinib_eye_disease
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Uveitis; Scleritis
MeSH Terms: conditions — Uveitis; Scleritis | interventions — tofacitinib; 5-(tetradecyloxy)-2-furancarboxylic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tofacitinib Treatment (Experimental): 11mg extended-release tofacitinib, once daily, oral
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: tofacitinib — tofacitinib extended release, 11mg, daily, oral
  Other Names: TOFA

SUMMARY:
Non-infectious inflammatory eye disease, such as uveitis and scleritis, is a chronic, auto-immune process that leads to vision loss. While steroids are effective in the short term, the side-effect profile of chronic steroid use necessitates the identification of effective steroid-sparing therapies. Tofacitinib is a small molecule that inhibits the signaling pathways of multiple inflammatory cytokines. The investigators plan to evaluate whether tofacitinib may have efficacy for patients with uveitis and / or scleritis.

DETAILED DESCRIPTION:
This study is a prospective, single-site, open-label investigation of tofacitinib for refractory uveitis. The study will be for 24 weeks, with potential 1-year extension for treatment responders. The patients will self-administer the medication.

Eligible patients would be those patients with a diagnosis of uveitis who meet the following criteria:

1. Disease sufficiently severe to require treatment with systemic corticosteroids, and
2. Referred from Ophthalmology to Rheumatology or Uveitis specialist for a steroid-sparing agent

For patients naive to oral steroid-sparing therapy (e.g., methotrexate, azathioprine, or mycophenolate), tofacitinib will be initiated as monotherapy. For patients who have failed or had only a partial response to oral steroid-sparing therapy, tofacitinib will be initiated as an add-on therapy. For patients intolerant to a conventional agent, tofacitinib will be initiated as replacement monotherapy. For patients who have failed biologic therapy (e.g. adalimumab), biologic therapy will be discontinued and tofacitinib will be initiated as replacement therapy without change to concurrent conventional steroid-sparing agents. Study visits will occur at baseline/enrollment, and weeks 4, 8, 12, 16, & 24 (+/- 2 weeks). Clinic visits may occur more frequently as determined by the treating physician. Laboratory monitoring (Table 1) will be obtained according to standard of care for drug toxicity monitoring. Clinical responses will be evaluated at 24 weeks, with the primary outcome defined as treatment failure.

All patients will undergo a predetermined oral steroid taper starting at 60mg of prednisone (or equivalent) and tapering over 14 weeks (Table 2). All patients will undergo a predetermined topical steroid drop taper starting at their current dose (Table 3).

Patients will have an ophthalmological evaluation by their treating ophthalmologist at Washington University. Steroid sparing therapy will be managed by rheumatologists or uveitis specialists at Washington University. All patients will be evaluated for an associated systemic rheumatologic condition.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of uveitis
* a clinical response to steroids
* active disease requiring at least 10mg of prednisone daily (or steroid equivalent)

Exclusion Criteria:

* suspected or confirmed ocular infection
* chronic or recurring infections, such as HIV
* renal insufficiency that would preclude safe administration of tofacitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2021-04-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Hassman, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Active uveitis despite at least 10mg prednisone for 2 weeks.
Period: Overall Study
Arm/Group | Tofacitinib Treatment
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Tofacitinib: single arm- tofacitinib 11mg daily
Arm/Group | Tofacitinib
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 58.8 [49 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure (Composite Outcome)
Description: new inflammatory lesions relative to baseline OR 2-step increase in anterior chamber cell or vitreous haze OR worsening of visual acuity by two or more rows on ETDRS chart
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Treatment
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Tofacitinib Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib Treatment (N=5)
cutaneous melanoma (Skin and subcutaneous tissue disorders) | 1 (1) — right upper extremity melanoma, with negative sentinel lymph nodes
squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) — squamous cell carcinoma on arm, fast-growing, history of multiple squamous cell carcinomas removed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03580343/Prot_SAP_000.pdf